CLINICAL TRIAL: NCT05644730
Title: Demonstration of an Artificial Intelligence Based Closed Loop Glucose Control System as a Therapeutic Modality in Type 1 and Type 2 Diabetic Patients
Brief Title: Closed Loop Glucose Control in Patients With Type 1 and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ideal Medical Technologies (Industry)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMT 2022-1_Version 1.0.7
Record Dates: First submitted 2022-11-17; First posted 2022-12-09 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Closed Loop Glucose Control; Artificial Pancreas; Artificial Intelligence; Glucose; Intensive Care Unit
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Early feasibility safety study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FUSION closed loop glucose control system safety study (Experimental): All subjects will be treated with the FUSION closed loop glucose control system for up to 24 hours
  Interventions: Device: Fusion closed loop glucose control system

INTERVENTIONS:
Device: Fusion closed loop glucose control system — The FUSION system will be used to control the subjects glucose to a range of 100-140 mg/dL. Data will be collected for up to 24 hours, or upon early termination of the study session.

SUMMARY:
This is a proof of concept safety study of an artificial intelligence based closed loop glucose control system designed for use in the intensive care unit setting.

The type 1 and type 2 diabetic subjects in this study will have their glucose controlled to a range of 100-140 mg/dL by a novel artificial intelligence based closed loop glucose control system for a period of 24 hours. The subjects will consume three standardized meals during the 24 hour study period.

DETAILED DESCRIPTION:
Tight glucose control in the intensive care unit (ICU) setting is difficult to achieve. The investigators hypothesize that a closed loop glucose control system based on artificial intelligence (AI) will improve upon the glucose control currently achieved by the current open loop manual methods, and that this improved glucose control may improve the outcomes of critically ill patients, including those with COVID-19.

This Earl Feasibility Study will test the ability of a prototype artificial intelligence based closed loop glucose control system named FUSION, to provide safe and effective glucose control in subjects with type 1 and type 2 diabetes in a clinical research center (CRC) setting. Subjects with type 1 diabetes have been chosen as safe and effective glucose control is difficult to achieve in these subjects during meal challenges. Subjects with type 2 diabetes have been chosen as they are insulin resistant, which makes their insulin resistance profile similar to that of ICU patients. As this is the first in human study of a new medical device, the controlled environment of the CRC is preferable to the less controlled environment of an ICU setting.

The prototype FUSION system to be used in this study will consist to two Dexcom G6 continuous glucose monitors (CGM), the AI-based glucose control software run on an all-in-one medical computer, and two syringe pumps. The prototype system is housed on a medical cart. Based on the average glucose value of the two Dexcom G6 CGM's, and the rules of the FUSION systems AI-based glucose control software, the FUSION system will make rate adjustments every 5-10 minutes to the intravenous infusion rates of short acting insulin (NovoLog) and dextrose (D10NS) under its control, in an attempt to keep the subjects glucose in the range of 100-140 mg/dL. The FUSION system only requires entry of the subjects study identification number and weight in kilograms to initiate the system.

For safety reasons, the subjects will have their blood glucose independently measured every 10-60 minutes on the point of care Nova StatStrip system, throughout the 24 hour study period.

The study has halting criteria to avoid recurrent instances of severe hypoglycemia (< 54 mg/dL).

The average of the two CGM's, that is used by the FUSION system for glucose control, will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18-70 years of age, inclusive.
2. Can understand and sign an informed consent, communicate with the investigator, and understand and comply with the protocol requirements.
3. Have had a diagnosis of type 1 or type 2 diabetes for a period of at least 1 year.
4. Use insulin injections at home for glucose control and are on a stable insulin regimen without more than a 20% change in their total daily insulin dose during the previous 3 months. Their total daily insulin dose during the previous 3 months will be confirmed through a review of the subject's electronic health record, insulin prescriptions, and insulin pump settings (if applicable).
5. Have a hemoglobin A1c (HbA1c) in the range of 7.0 - 10.0%.
6. Have a hemoglobin in the normal range for sex:

   1. Females: 12-15.5 grams/dL.
   2. Males: 13.5-17.5 grams/dl.
7. Have adequate venous access sites in upper extremities.
8. Body weight between 40 - 150 kg.

Exclusion Criteria:

1. Have participated in an interventional medical, surgical, or pharmaceutical study within 30 days of screening.
2. Have a known hypersensitivity to any of the components of study treatment.
3. Have skin disease/injury at Dexcom G6 CGM insertion site(s) that would prevent insertion of the CGM.
4. Currently abuses drugs or alcohol or has a history of abuse that in the investigator's opinion would cause the individual to be noncompliant.
5. Have a medical condition that in the opinion of the investigator could affect study participation and/or personal well-being.
6. Have a clinically significant history or presence of any of the following conditions:

   1. Hepatic failure or has alanine aminotransferase (ALT) greater than 3 times the upper limit of normal.
   2. Has an estimated glomerular filtration rate (GFR) <60 ml/min/1.73 m2 or End Stage Kidney Disease on renal replacement therapy.
   3. Type 2 diabetic subjects who have a C-peptide level less than 0.2 nmol/L (these subjects will be referred to their primary care doctor or endocrinologist for further work up).
   4. Have congestive heart failure of class 1 or greater on the New York Heart Association (NYHA) classification system.
   5. Have a history of seizures.
   6. Have a history of cerebrovascular accident.
   7. Have a history of ischemic heart disease.
7. For female subjects of potential childbearing age (age 18 to 55) they will be excluded if:

   1. Pregnant.
   2. Refuse to agree to a pregnancy test at the time of enrollment.
   3. Have a positive urine pregnancy test at the time of enrollment.
8. Have a positive COVID-19 test within 14 days of visit 3.
9. Have any COVID-19 related symptoms in the 14-day period prior to visit 3.
10. Have a known unprotected COVID-19 exposure in the 14-day period prior to visit 3.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon DeJournett, MD, Study Director — Ideal Medical Technologies; Francisco Pasquel, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeJournett L, DeJournett J. In Silico Testing of an Artificial-Intelligence-Based Artificial Pancreas Designed for Use in the Intensive Care Unit Setting. J Diabetes Sci Technol. 2016 Nov 1;10(6):1360-1371. doi: 10.1177/1932296816653967. Print 2016 Nov. PMID 27301982
- [Background] DeJournett J, DeJournett L. Comparative Simulation Study of Glucose Control Methods Designed for Use in the Intensive Care Unit Setting via a Novel Controller Scoring Metric. J Diabetes Sci Technol. 2017 Nov;11(6):1207-1217. doi: 10.1177/1932296817711297. Epub 2017 Jun 22. PMID 28637358
- [Background] DeJournett J, Nekludov M, DeJournett L, Wallin M. Performance of a closed-loop glucose control system, comprising a continuous glucose monitoring system and an AI-based controller in swine during severe hypo- and hyperglycemic provocations. J Clin Monit Comput. 2021 Apr;35(2):317-325. doi: 10.1007/s10877-020-00474-2. Epub 2020 Jan 31. PMID 32006145
- [Background] DeJournett L. Essential elements of the native glucoregulatory system, which, if appreciated, may help improve the function of glucose controllers in the intensive care unit setting. J Diabetes Sci Technol. 2010 Jan 1;4(1):190-8. doi: 10.1177/193229681000400124. PMID 20167184
- [Background] Sardu C, D'Onofrio N, Balestrieri ML, Barbieri M, Rizzo MR, Messina V, Maggi P, Coppola N, Paolisso G, Marfella R. Outcomes in Patients With Hyperglycemia Affected by COVID-19: Can We Do More on Glycemic Control? Diabetes Care. 2020 Jul;43(7):1408-1415. doi: 10.2337/dc20-0723. Epub 2020 May 19. PMID 32430456

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Outcome
Description: Percent of All Glucose Values Within Glucose Range < 70 mg/dL
Time Frame: From beginning of use of the FUSION System to end of use of the FUSION System, which will be a period of time up to 24 hours
Measure: Mean (Standard Deviation); unit: Percentage of all glucose values
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Percentage of all glucose values | 1.4 (2.7)

2. Primary Outcome: Primary Efficacy Outcome
Description: Percent of All Glucose Values Within Glucose Range 70-180 mg/dL
Time Frame: From beginning of use of FUSION System to end of use of FUSION System, which will be a period of time of up to 24 hours
Measure: Mean (Standard Deviation); unit: Percentage of all glucose values
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Percentage of all glucose values | 79.0 (21.3)

3. Secondary Outcome: Percent of All Glucose Values Within Glucose Range < 54 mg/dL
Description: The percentage of all glucose values that less than 54 mg/dL
Time Frame: From beginning of use of the FUSION System to end of use of the FUSION System, which will be a period of time of up to 24 hours
Measure: Mean (Standard Deviation); unit: Percentage of all glucose values
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Percentage of all glucose values | 0 (0)

4. Secondary Outcome: Percent of All Glucose Values Within Glucose Range > 180 mg/dL
Description: Percentage of all glucose values that are greater than 180 mg/dL
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of all glucose values
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Percentage of all glucose values | 19.6 (22.0)

5. Secondary Outcome: Percent of All Glucose Values Within Glucose Range > 250 mg/dL
Description: The percentage of all glucose values that are greater than 250 mg/dL
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of all glucose values
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Percentage of all glucose values | 2.9 (4.4)

6. Secondary Outcome: Average Glucose Value in mg/dL
Description: The average of all measured glucose values in mg/dL
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
mg/dL | 148.4 (25.1)

7. Secondary Outcome: Percent Coefficient of Variation of Glucose
Description: The percent coefficient of variation of glucose will be calculated by dividing the standard deviation of the average glucose value in mg/dL by the average glucose value in mg/dL, then multiplying this value by 100
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Coefficient of Variation
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Percentage of Coefficient of Variation | 21.3 (5.3)

8. Secondary Outcome: Weight in Kilograms
Description: Average weight in kilograms of the subjects
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Kilograms | 88.2 (14.7)

9. Secondary Outcome: Body Mass Index
Description: The body mass index was calculated by dividing the subjects weight in kilograms by their height in meters squared
Time Frame: As measured at the start of the closed loop glucose control session
Measure: Mean (Standard Deviation); unit: Kilograms/Height in meters squared
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Kilograms/Height in meters squared | 31.0 (6.1)

10. Secondary Outcome: Total Daily Dose of Insulin in Units/Kilogram
Description: The subjects total daily dose of insulin used prior to the start of the closed loop glucose control session was calculated by adding up all of the insulin doses used by the subjects (both short and long acting insulin) in units and dividing this value by the subjects weight in Kilograms
Time Frame: As measured prior to the start of the closed loop glucose control session
Measure: Mean (Standard Deviation); unit: Units Insulin/Kilogram per day
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Units Insulin/Kilogram per day | 0.9 (0.4)

11. Secondary Outcome: Hemoglobin A1c Percentage Level
Description: The subjects hemoglobin A1c measurement from a blood draw taken within 2 weeks of the start of the closed loop glucose control session
Time Frame: As measured within 2 weeks of the start of the closed loop glucose control session
Measure: Mean (Standard Deviation); unit: Percentage of glycated hemoglobin
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
Percentage of glycated hemoglobin | 8.5 (0.8)

12. Secondary Outcome: C-Peptide Level in ng/mL
Description: C-Peptide level as measured from a blood draw
Time Frame: As measured from a blood draw taken within 2 weeks of the start of the closed loop glucose control session
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
Number analyzed (Participants) | 7
ng/mL | 1.5 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the closed loop glucose control session, which was a period of time of up to 24 hours for each subject
Description: The following guidelines were used to describe adverse event severity:
  * Mild - Events require minimal or no treatment and do not interfere with the participant's daily activities.
  * Moderate - Events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning.
  * Severe - Events interrupt a participant's usual daily activity and may require systemic drug therapy or other treatment.
Arm/Group | FUSION Closed Loop Glucose Control System Safety Study
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FUSION Closed Loop Glucose Control System Safety Study (N=7)
Sustained Glucose Value > 250 mg/dL (Endocrine disorders) | 1 (1) — Subjects with a sustained glucose value > 250 mg/dL for a period of time of greater than or equal to 60 minutes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT05644730/Prot_SAP_000.pdf